CLINICAL TRIAL: NCT07338513
Title: User-centric Study of Patients' Receptiveness Towards the Web-based Automated Vision Impairment Gaze-tracking Analysis Systems
Acronym: AVIGA-SURVEY
Status: Not yet recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Laude Augustinus, Senior Consultant, Tan Tock Seng Hospital
Other Study IDs: 2025-1535
Record Dates: First submitted 2025-11-20; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: user interface; user experience; Technology Acceptance Model; System Usability Scale
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Age-Related Macular Degeneration (AMD) is the leading cause of central vision loss among older adults worldwide. Patients with AMD often require frequent monitoring of visual function and disease progression, typically through multiple follow-up visits involving optical coherence tomography (OCT), visual acuity testing (VA), and clinical consultations.

While digital self-monitoring tools have emerged as promising solutions to reduce the burden of in-clinic visits, many elderly patients face challenges in engaging with these platforms due to visual impairment, limited digital literacy, and poorly optimised user interfaces. These barriers may reduce patient willingness to adopt such systems and undermine their long-term effectiveness.

To address this gap, the study team has developed the web-based AVIGA (Automated Vision Impairment Gaze-tracking Analysis) system, which is a portable, self-administered, home-based digital monitoring system designed to minimise cognitive load and maximise usability for elderly AMD patients. The platform integrates patient-centred design principles such as simplified navigation, optimised text, and multimodal feedback (visual and audio) to empower users to independently track their visual health.

A prospective, single-site usability trial to evaluate the AVIGA platform using validated human factors measures: the System Usability Scale (SUS), the Technology Acceptance Model (TAM) will be conducted. By examining the relationship between usability, cognitive load, and perceived empowerment, this study aims to identify critical user interface and user experience (UI/UX) design factors that influence willingness to adopt and sustain use of digital health tools among elderly AMD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in the age group ≥ 55 to 99 years old.
2. Both genders
3. Able to understand verbal spoken instructions in British/American English, Chinese or Bahasa Melayu and demonstrate device functionality and implementation.
4. Subjects undergoing treatment for Wet-AMD without any signs and symptoms of recurrence of active AMD (AMD recurrence: choroidal neovascularisation, intraretinal or subretinal fluid is present) with OCT lesion fluid volume more than 2mm2 or ILM height more than 300µm.
5. Ability to comply with the study protocol, in the investigator's judgment.
6. Subjects must be able to understand and provide informed consent. A signed informed consent form must be provided before any study assessments.

Exclusion Criteria:

1. Unable to understand verbal spoken instructions and demonstrate device functionality and implementation.
2. Unable to turn on and connect their computer to the AVIGA platform independently.
3. Any ocular surgery in the previous 3 months, or vitrectomy in the previous 12 months
4. Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye
5. Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
6. Any prior or concomitant treatment for CNV or vitreomacular-interface abnormalities in the study eye.
7. History of idiopathic or autoimmune-associated uveitis in either eye
8. Active ocular inflammation or suspected or active ocular or periocular infection in either eye.
9. Severe cognitive impairment, comorbid conditions severely limiting participation (e.g., advanced hearing loss)

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously recruited with recurrent vision problems diagnosed with active Wet-AMD at the TTSH Specialist Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assess System Usability | Baseline, Mid-point (6 months from baseline ±3 months), End-point (12 months from baseline ±3 months)
  Measure and evaluate overall system usability across three checkpoints (Baseline, Mid-point, and End-point) using the System Usability Scale (SUS), a 10-item questionnaire rated on a 5-point Likert scale.
Assess System Acceptance | Baseline, Mid-point (6 months from baseline ±3 months), End-point (12 months from baseline ±3 months)
  Measure and evaluate overall acceptance towards system adoption across three checkpoints (Baseline, Mid-point, and End-point) using 8 items from the Technology Acceptance Model (TAM), rated on a 5-point Likert scale.

SECONDARY OUTCOMES:
Track Change Over Time | Baseline, Mid-point (6 months from baseline ±3 months), End-point (12 months from baseline ±3 months)
  Compare the changes in expectation (Baseline) versus lived experience (Mid-point, End-point) scores taken from the combined SUS and TAM to identify how usability perceptions and adoption intentions evolve with continued use.

CONTACTS AND LOCATIONS:
Overall Officials: Augustinus Laude, MBChB, Principal Investigator — Tan Tock Seng Hospital; Zheng Kuang Noel Soh, BSc, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

REFERENCES:
- [Background] Huiying Liu, Wong D, Ai Ping Yow, Yanwu Xu, Fengshou Yin, Laude A, Tock Han Lim. Determining the difference in eyegaze measurements in individuals with age related macular degeneration. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:1348-1351. doi: 10.1109/EMBC.2016.7590957. PMID 28268575
- [Background] Huiying Liu, Yanwu Xu, Damon Wong, Ai Ping Yow, Laude A, Tock Han Lim. Detecting impaired vision caused by AMD from gaze data. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:3142-3145. doi: 10.1109/EMBC.2017.8037523. PMID 29060564
- [Background] Liu, H., et al., Vision assessment based on gaze. 2019, AGENCY FOR SCIENCE, TECHNOLOGY AND RESEARCH [SG/SG]; 1 Fusionopolis Way, #20-10 Connexis North Tower, Singapore 138632, SG: Singapore.
- [Background] Goldberg, J.H. and X.P. Kotval, Computer interface evaluation using eye movements: methods and constructs. International journal of industrial ergonomics, 1999. 24(6): p. 631-645.
- [Background] Loewenstein A; Richard & Hinda Rosenthal Foundation. The significance of early detection of age-related macular degeneration: Richard & Hinda Rosenthal Foundation lecture, The Macula Society 29th annual meeting. Retina. 2007 Sep;27(7):873-8. doi: 10.1097/IAE.0b013e318050d2ec. PMID 17891011
- [Background] Goldberg, J.H. and A.M. Wichansky, Eye tracking in usability evaluation: A practitioner's guide, in the Mind's Eye. 2003, Elsevier. p. 493-516.
- [Background] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study (AREDS): design implications. AREDS report no. 1. Control Clin Trials. 1999 Dec;20(6):573-600. doi: 10.1016/s0197-2456(99)00031-8. PMID 10588299
- [Background] Chew EY, Clemons TE, Agron E, Sperduto RD, Sangiovanni JP, Davis MD, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Ten-year follow-up of age-related macular degeneration in the age-related eye disease study: AREDS report no. 36. JAMA Ophthalmol. 2014 Mar;132(3):272-7. doi: 10.1001/jamaophthalmol.2013.6636. PMID 24385141
- [Background] AREDS2 Research Group; Chew EY, Clemons T, SanGiovanni JP, Danis R, Domalpally A, McBee W, Sperduto R, Ferris FL. The Age-Related Eye Disease Study 2 (AREDS2): study design and baseline characteristics (AREDS2 report number 1). Ophthalmology. 2012 Nov;119(11):2282-9. doi: 10.1016/j.ophtha.2012.05.027. Epub 2012 Jul 26. PMID 22840421
- [Background] AREDS2-HOME Study Research Group; Chew EY, Clemons TE, Bressler SB, Elman MJ, Danis RP, Domalpally A, Heier JS, Kim JE, Garfinkel R. Randomized trial of a home monitoring system for early detection of choroidal neovascularization home monitoring of the Eye (HOME) study. Ophthalmology. 2014 Feb;121(2):535-44. doi: 10.1016/j.ophtha.2013.10.027. Epub 2013 Nov 8. PMID 24211172
- [Background] Mathew R, Sivaprasad S. Environmental Amsler test as a monitoring tool for retreatment with ranibizumab for neovascular age-related macular degeneration. Eye (Lond). 2012 Mar;26(3):389-93. doi: 10.1038/eye.2011.326. Epub 2011 Dec 16. PMID 22173073
- [Background] Ai Ping Yow, Damon Wong, Huiying Liu, Hongyuan Zhu, Ivy Jing-Wen Ong, Laude A, Tock Han Lim. Automatic visual impairment detection system for age-related eye diseases through gaze analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:2450-2453. doi: 10.1109/EMBC.2017.8037352. PMID 29060394
- [Background] Trevino R, Kynn MG. Macular function surveillance revisited. Optometry. 2008 Jul;79(7):397-403. doi: 10.1016/j.optm.2007.09.017. PMID 18577497
- [Background] Kawasaki R, Wang JJ, Aung T, Tan DT, Mitchell P, Sandar M, Saw SM, Wong TY; Singapore Malay Eye Study Group. Prevalence of age-related macular degeneration in a Malay population: the Singapore Malay Eye Study. Ophthalmology. 2008 Oct;115(10):1735-41. doi: 10.1016/j.ophtha.2008.02.012. Epub 2008 Apr 25. PMID 18439679
- [Background] Brooke, John.
- [Background] Davis, Fred D.